CLINICAL TRIAL: NCT06939023
Title: Laparoscopic Versus Robot-assisted Left-sided Pancreatectomy for Benign and Pre-malignant Lesions (DIPLOMA-3): an International Multicenter Patient-blinded Randomized Controlled Trial
Brief Title: Laparoscopic Versus Robot-assisted Left-sided Pancreatectomy for Benign and Pre-malignant Lesions (DIPLOMA-3)
Acronym: DIPLOMA-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Erasmus Medical Center (Other); Medisch Spectrum Twente (Other); Maastricht University Medical Center (Other); University Medical Center Groningen (Other); Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, M.G. Besselink, prof. dr. M.G. Besselink, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL88413.018.24
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pancreatectomy; Distal Pancreatectomy (DP); Pancreatic Neoplasms; Pancreatic Adenoma; Pancreatic Cyst; Pancreatic Cystadenoma; Surgery; Minimally Invasive Surgical Technique; Minimally Invasive Distal Pancreatectomy; Minimally Invasive Surgery
Keywords: pancreas surgery; left-sided pancreatectomy; distal pancreatectomy; minimally invasive surgery; robot-assisted pancreatectomy; left pancreatectomy; robotic pancreatectomy; laparoscopic pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic adenoma; Pancreatic Cyst

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient-blinded up to post-operative day 5. Blinded adjudication committee assessing the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic minimally invasive left-sided pancreatecomy (Active Comparator): Laparoscopic minimally invasive left-sided pancreatecomy
  Interventions: Procedure: Laparoscopic minimally invasive left-sided pancreatecomy
- Robot-assisted minimally invasive left-sided pancreatecomy (Experimental): Robot-assisted minimally invasive left-sided pancreatecomy
  Interventions: Procedure: Robot-assisted minimally invasive left-sided pancreatecomy

INTERVENTIONS:
Procedure: Laparoscopic minimally invasive left-sided pancreatecomy — Laparoscopic minimally invasive left-sided pancreatecomy
  Arms: Laparoscopic minimally invasive left-sided pancreatecomy
Procedure: Robot-assisted minimally invasive left-sided pancreatecomy — Robot-assisted minimally invasive left-sided pancreatecomy
  Arms: Robot-assisted minimally invasive left-sided pancreatecomy

SUMMARY:
The DIPLOMA-3 trial is an international, multicenter, patient-blinded randomized controlled trial comparing laparoscopic and robot-assisted left-sided pancreatectomy. Patients with an indication for elective left-sided pancreatecomy for benign or premalignant lesions in the body or tail of the pancreas and considered eligible will be randomized between laparoscopic and robot-assisted resection.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years;
* Indication for elective left-sided pancreatectomy, either spleen-preserving or non-preserving (because of proven or suspected left-sided benign or premalignant disease);
* Both robot-assisted and laparoscopic left-sided pancreatectomy are technically feasible for resection, according to the local treatment team;
* Fit to undergo left-sided pancreatectomy according to the surgeon and anaesthesiologist;
* Written informed consent

Exclusion Criteria:

* Suspected pancreatic ductal adenocarcinoma;
* Tumor or cyst larger than 8 cm;
* Required resection or ablation of organs other than pancreas and spleen;
* Tumor involvement or abutment of major vessels (celiac trunk, mesenteric artery or vena cava);
* Pregnancy;
* Body mass index >40 kg/m2;
* Participation in another study with interference of study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
COMPOS-panc left score | 90 days
  The COMPOS-panc left score is a recently developed, severity-weighted composite outcome measure for pancreatic surgery. It combines perioperative and postoperative outcomes into a single composite outcome measure. This score includes the following parameters, measured at 90-days postoperative: unplanned blood transfusion, emergency conversion to open surgery, postoperative pancreatic fistula (POPF), postpancreatectomy hemorrhage (PPH), other complications requiring intervention, multi-organ failure, mortality, length of hospital stay and readmission requiring intervention.

SECONDARY OUTCOMES:
Total hospital-related costs | 90 days
  To examine total hospital-related costs, the following costs will be considered up to 90 days postoperative:
  1. Direct cost of the operation
  2. Direct cost of the post-operative hospital stay
  3. Direct cost of follow-up period, including readmission, outpatient visits, emergency room visits and reintervention
Spleen-preservation rate and spleen-preservation technique | Surgery
  Compare L-MILP and R-MILP for spleen-preservation rate and spleen-reservation technique (Kimura versus Warshaw technique)
Pancreatic surgery specific complications | 90 days
  Complications including pancreatic fistula, delayed gastric emptying, postoperative bleeding, wound infection, other gastrointestinal leakage, re-interventions (radiographic, endoscopic, surgical), ICU admission, in hospital, 30- and 90-day mortality.

OTHER OUTCOMES:
Operative outcomes | Surgery
  Total operative time (first skin incision to fully closed skin incisions, min.); Time of reconstruction phase; Estimated intraoperative blood loss (mL); Serious intraoperative complications; Conversion; Reason for conversion; Surgeon's mental strain (measured at the end of surgery).
Length of hospital stay | 90 days postoperatively
  Days from surgery to discharge; Readmission rates; Total of hospitalized days.
Patient-reported outcomes | 1 year postoperative
  (Health-related) Quality of Life measurement using validated EORTC questionnaires: Baseline, 1-, 3-, 6- months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Mohammad Abu Hilal, MD PhD, Principal Investigator — University of Jordan; Prof. Marc Besselink, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands